CLINICAL TRIAL: NCT00002647
Title: Photodynamic Therapy For Childhood Brain Tumors, A Phase I Study
Brief Title: Photodynamic Therapy With Porfimer Sodium in Treating Patients With Refractory Brain Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical College of Wisconsin (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000064165; MCW-7594; MCW-CHW-511; MCW-CHW-9411; NCI-V95-0652
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2009-06

CONDITIONS: Brain and Central Nervous System Tumors; Metastatic Cancer
Keywords: recurrent adult brain tumor; tumors metastatic to brain; recurrent childhood brain stem glioma; recurrent childhood anaplastic astrocytoma; recurrent childhood anaplastic oligoastrocytoma; recurrent childhood anaplastic oligodendroglioma; recurrent childhood cerebellar astrocytoma; recurrent childhood cerebral astrocytoma; recurrent childhood diffuse astrocytoma; recurrent childhood fibrillary astrocytoma; recurrent childhood gemistocytic astrocytoma; recurrent childhood giant cell glioblastoma; recurrent childhood glioblastoma; recurrent childhood gliomatosis cerebri; recurrent childhood gliosarcoma; recurrent childhood oligodendroglioma; recurrent childhood pilocytic astrocytoma; recurrent childhood pilomyxoid astrocytoma; recurrent childhood pleomorphic xanthoastrocytoma; recurrent childhood protoplasmic astrocytoma; recurrent childhood subependymal giant cell astrocytoma; recurrent childhood visual pathway and hypothalamic glioma; recurrent childhood visual pathway glioma; recurrent childhood pineoblastoma; recurrent childhood supratentorial primitive neuroectodermal tumor; recurrent childhood medulloblastoma; recurrent childhood ependymoma; recurrent childhood brain tumor; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult anaplastic meningioma; adult anaplastic oligodendroglioma; adult brain stem glioma; adult central nervous system germ cell tumor; adult choroid plexus tumor; adult craniopharyngioma; adult diffuse astrocytoma; adult ependymoblastoma; adult ependymoma; adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma; adult medulloblastoma; meningeal melanocytoma; adult meningeal hemangiopericytoma; adult oligodendroglioma; adult papillary meningioma; adult pilocytic astrocytoma; adult pineal gland astrocytoma; adult pineoblastoma; adult pineocytoma; adult subependymal giant cell astrocytoma; adult subependymoma; adult supratentorial primitive neuroectodermal tumor (PNET); childhood grade I meningioma; childhood grade II meningioma; childhood grade III meningioma; adult grade III meningioma; childhood central nervous system germ cell tumor; childhood choroid plexus tumor; childhood craniopharyngioma; childhood infratentorial ependymoma; childhood supratentorial ependymoma; childhood low-grade cerebral astrocytoma; childhood high-grade cerebral astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Neoplasm Metastasis; Brain Neoplasms; Astrocytoma; Oligodendroglioma; Glioblastoma; Neoplasms, Neuroepithelial; Optic Nerve Glioma; Medulloblastoma; Familial ependymoma; Ependymoma; Meningioma; Choroid Plexus Neoplasms; Craniopharyngioma; Neuroectodermal Tumors, Primitive; Gliosarcoma; Pinealoma; Glioma, Subependymal | interventions — Verteporfin

INTERVENTIONS:
Drug: verteporfin
Procedure: conventional surgery

SUMMARY:
RATIONALE: Photodynamic therapy uses light and photosensitizing drugs to kill tumor cells and may be an effective treatment for refractory brain tumors.

PURPOSE: This phase I trial is studying the side effects and best dose of photodynamic therapy using porfimer sodium in treating patients with refractory brain tumors, including astrocytoma, ependymoma, and medulloblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose of benzoporphyrin monoacid ring A in patients with refractory brain tumors undergoing cavitary photoillumination photodynamic therapy.
* Determine the effect of this regimen on neurotoxicity, clinical state, imaging changes, and survival of these patients.

OUTLINE: This is a dose-escalation study. Patients are stratified according to tumor location (posterior fossa tumors vs all other brain tumors).

Patients receive benzoporphyrin monoacid ring A (BPD-MA) IV preoperatively. Approximately 3 hours after BPD-MA administration, patients undergo craniotomy with photoillumination of the tumor. Patients with tumors greater than 2 cm in diameter also undergo gross tumor resection.

Cohorts of 3-6 patients receive escalating doses of BPD-MA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose immediately preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Three additional patients are treated at the MTD.

Patients are followed at 4 and 6 weeks, every 3 months for 1 year, every 6 months for 1 year, and then annually thereafter.

PROJECTED ACCRUAL: A minimum of 24 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of supratentorial or infratentorial brain tumor

  * Localized, non-disseminated
  * Primary tumor or solitary metastasis
  * Recurrent or progressive
  * Unresectable
  * Negative CSF
* Must have failed standard therapy including radiotherapy
* Measurable disease as evidenced by CT scan or MRI

  * Single or multiple masses accessible to light administration

PATIENT CHARACTERISTICS:

Age:

* 3 to 70

Performance status:

* Not specified

Life expectancy:

* At least 2 months

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm3
* May transfuse platelets

Hepatic:

* PT and PTT normal

Renal:

* Not specified

Other:

* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 6 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior brachytherapy

Surgery:

* See Disease Characteristics

Other:

* No other concurrent antitumor therapy

Ages: 3 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 1994-05

CONTACTS AND LOCATIONS:
Overall Officials: Harry T. Whelan, MD, Study Chair — Medical College of Wisconsin
Locations (2):
- United States (2):
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Background] Schmidt MH, Bajic DM, Reichert KW 2nd, Martin TS, Meyer GA, Whelan HT. Light-emitting diodes as a light source for intraoperative photodynamic therapy. Neurosurgery. 1996 Mar;38(3):552-6; discussion 556-7. doi: 10.1097/00006123-199603000-00025. PMID 8837808